CLINICAL TRIAL: NCT03660423
Title: The Effects of Dance Training on Postural Stability in Adults With Developmental Disabilities
Brief Title: Dance Training for Developmental Disabilities
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to COVID-19 and decreased ability to safely dance in person
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1804-717
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Developmental Disability
Keywords: Dance
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance Group (Experimental): Dance group will participate in a 60 minute integrative dance class two times per week
  Interventions: Other: Integrative Dance
- Control Group (No Intervention): The Control group will continue with normal activities, not participating in the dance intervention.

INTERVENTIONS:
Other: Integrative Dance — Integrative dance may be defined as dance that encourages the participation of all individuals, regardless of ability, supporting and celebrating these differences as a community. In the intervention, adults with developmental disabilities will be dancing in a contemporary dance class alongside college students.
  Arms: Dance Group

SUMMARY:
the purpose of this current study is to examine the changes in postural stability in adult individuals with developmental disabilities following exposure to a college based integrative dance training course. Integrative dance may be defined as dance that encourages the participation of all individuals, regardless of ability, supporting and celebrating these differences as a community. It is hypothesized that a significantly reduced body sway will be observed in participants following a college based integrative dance training course. Furthermore, in participants that continue dancing in the program over multiple semesters, it is hypothesized that there will be an inverse relationship between body sway and dance participation over time (IE: As participants dance more, body sway will continue to decrease).

DETAILED DESCRIPTION:
11. Procedures:

11.1 Bridges to Skidmore Course Information DA209, Bridges to Skidmore: The Dance Experience class will be held twice per week in the dance facilities or Tang teaching museum. This course will be taught by Dr. Sarah DiPasquale who will also lead the dance class sessions each week. Dependent on space constraints and learning goals each semester, the class will convene in the dance studios, dance theater, Tang teaching museum or intramural gym of the Williamson Sports Center. The Williamson Sports Center and Tang museum are accessible buildings with multiple handicap accessible parking spots available for the Saratoga Bridges staff to transport participants. Each week the participants will partake in 100-120 minutes of contemporary dance training; participants work up to a 30 minute warm up period at the beginning of class and then take a short break to get a drink or use the bathroom. Chairs are also set up on all sides of the room so individuals can rest or take a break if they wish. They will learn the basic positions and combinations used in Contemporary Dance, including: Plié, Tendu, Degagé, Rond de Jambe, Frappé, Chassé, Sauté, Pas de Bourrée, Glissade, and Révérance. Additional Contemporary Dance movements and patterns will be employed utilizing a mixture of fall and recovery techniques consistent with this discipline's movement vocabulary. A minimum of two staff members from Saratoga Bridges will be in attendance during the class period in addition to the 8-10 students helping with the class. If a participant chooses not to dance for the full duration of a given class period, a Bridges staff member will assist them out of the studio to wait comfortably in the lobby of the dance center, dance gym or sports center until the class ends and their transportation arrives. A staff member from Saratoga Bridges will remain with the participant outside of the dance studio. They may also rejoin the class at any time, should they choose.

Skidmore dance students will register for a 1-credit course through the dance department entitled Bridges to Skidmore: The Dance Experience (DA271-001). Skidmore students registered in this class will be matched with a cohort of Bridges participants (ideally a 4:1 ratio or less). These cohorts will work together in the classroom enabling each member to get to know one another throughout the duration of the semester. As the Bridges participants will come to class with a wide range of physical and intellectual abilities, the small group cohort embedded within the larger class setting will allow the student leaders to assist each person in a way that meets their individual learning and/or mobility needs.

Prior to any participation in Bridges to Skidmore: The Dance Experience, an intake form will be completed by a staff member at Saratoga Bridges. This staff member must be a health care provider who has full access to the participants protected health information (PHI).

The only person who will have full access to the completed intake forms will be Dr. Sarah DiPasquale PT, DPT. Student data collectors will have limited access to these files in order to input the information into the database. Prior to any student access to files containing PHI, the names of the participants will be removed from the documents and replaced with the participant ID numbers. Additionally, this access will be under direct faculty supervision and for only the amount of time needed to input the data. These files will be kept in a locked filing cabinet in office 228 of the Williamson Sports Center at all times and will not be removed from the office.

The first day of class for Bridges to Skidmore: The Dance Experience will be a training session for the Skidmore student cohort leaders. We will invite a member of the Saratoga Bridges medical or administrative team to talk with the class about working with people with DD. We will discuss appropriate interactions and confidentiality during the class.

*Please note: Student cohort leaders are not synonymous with student data collectors. Student cohort leaders will not have access to any data collected for the purposes of research. They will be participating only in the 1 credit dance course aspect of the Bridges to Skidmore: The Dance Experience project.

11.2 Data Collection Data collection will take place at the Saratoga Bridges facility, the multipurpose room (Williamson Sports Center) or the intramural gym (Williamson Sports Center) prior to the program commencement with post-testing to be completed the week of, or following, the final performance/graduation ceremony. Of great importance during data collection is the comprehension of the participants during the examination. While tests will be verbally explained/instructed, a physical demonstration of the measurement will be presented prior to administration. This will help to create clear expectations for the test (specifically for those with decreased abilities to comprehend complex verbal explanations), help to decrease any fear or anxiety surrounding the process, and potentially increase the reliably of test-retest procedures in this population.

Data collection will be overseen by Dr. Sarah DiPasquale and assisted by 2-3 student researchers from Skidmore College each semester. Student data collectors will be trained in all procedures and techniques directly by the supervising faculty members prior to any data collection and must be able to demonstrate competency in testing prior to administering any tests on participants.

Both the pre and post data collection will take approximately 15 minutes per participant at each testing session. Participants will receive instructions prior to each trial of 30 seconds and 2 researchers will always be present on either side of the participant should they lose their balance. Participants will be asked to stay in a static standing position for 3 trials of 30 seconds while standing on a Wii board in four of the following conditions : 1) bilateral stance with eyes open, 2) bilateral stance with eyes closed, 3) unilateral stance on the right limb 4) unilateral stance on the left limb 5) bilateral stance with eyes open on foam 6) bilateral stance with eyes closed on foam 7) unilateral stance on the right limb on foam and 8) unilateral stance on the left limb on foam. All three trials will happen back to back before moving on to the next condition. Different patterns of the four conditions will be utilized each year as research progresses although no more than four conditions will be utilized each semester as to minimize the time required of the participant for testing. Each semester, the participants will be tested under the same four conditions. Participants will be given a 15 seconds rest period between each trial and will be told they may rest at any moment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be registration in a Saratoga Bridges Day Habilitation program, being over the age of 18, and a statement from the physician in the participant's medical files at Bridges allowing unrestrictive activities.

Exclusion Criteria:

* Exclusion criteria will be active participation in a physical therapy program with the goal of improving functional mobility and participation in a consistent exercise class that has the potential to improve physical function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Body Sway | 12 weeks
  Body sway will be measured utilizing wii balance boards

CONTACTS AND LOCATIONS:
Overall Officials: Sarah DiPasquale, DPT, Principal Investigator — Skidmore College
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dipasquale S, Canter B, Roberts M. Integrative Dance for Adults with Down Syndrome: Effects on Postural Stability. Int J Exerc Sci. 2020 Sep 1;13(3):1317-1325. doi: 10.70252/FETH2009. eCollection 2020. PMID 33042366